CLINICAL TRIAL: NCT02975531
Title: Simulator of Pompage Technique for Education and Training of Physiotherapists
Brief Title: Simulator of Pompage Technique for Physiotherapists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Annie France Frère Slaets, PhD, University of Mogi das Cruzes
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 0121.0.237.00007
Record Dates: First submitted 2016-03-09; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Musculoskeletal Pain; Contracture
Keywords: Pompage
MeSH Terms: conditions — Musculoskeletal Pain; Contracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Simulator's construction (Experimental): To build the simulator was selected a volunteer (VF) as a model. This volunteer had no complaints of pain or trauma to the cervical region. This region was used to collect the displacement of the skin and cytometry neck.
  Interventions: Other: Simulator's construction
- Model Features (Experimental): Thirty-nine volunteers (GT) were selected men and women aged over 18 years without history of trauma in the cervical region in order to determine the characteristics of the model: skin elasticity and cirtometry neck.
  Interventions: Other: Model Features
- Parameterization technique (Experimental): Five physiotherapists (GP) with at least 5 years of experience in the technique were selected to perform the technique on the simulator and complete a questionnaire in order to evaluate the texture and skin elasticity, the curvature and size of the cervical spine format. They scored these items from the Likert scale. After evaluation they used the simulator to generate a standard guide training.
  Interventions: Other: Parameterization technique
- Simulator training (Experimental): Twenty-six volunteers (GE) were selected, men and women, aged over 18 years without prior knowledge of the technique for simulator training.
  Interventions: Other: Simulator training
- Training Evaluation (Experimental): A physical therapist (VE) was selected to evaluate the volunteers (GE) before and after training in the simulator.
  Interventions: Other: Training Evaluation

INTERVENTIONS:
Other: Simulator's construction — Model to build the mold for the simulator
  Other Names: VF
  Arms: Simulator's construction
Other: Model Features — Volunteers to determine the elasticity of the skin and cirtometry neck to compare with the simulator.
  Other Names: GT
  Arms: Model Features
Other: Parameterization technique — Evaluation of the simulator features and parameterization of the Pompage technique in the simulator.
  Other Names: GP
  Arms: Parameterization technique
Other: Simulator training — Training of pompage technique using the simulator.
  Other Names: GE
  Arms: Simulator training
Other: Training Evaluation — Evaluation of volunteers from GE group before and after training with the simulator.
  Other Names: VE
  Arms: Training Evaluation

SUMMARY:
Parameterize the Pompage technique with an anatomical model cervical region to simulate specific procedures. Quantify the times, displacements, and facilitate the training of students and professional of physical therapy.

DETAILED DESCRIPTION:
Manual techniques are taught and trained with practical demonstration without technology support to measure them, so they are difficult to reproduce. This difficulty increases in Pompage technique because the student is not able to estimate the displacement on the skin. In this research, to parameterize and train the technique was developed and validated an anatomical model of the cervical region, with silicone and latex rubber. The anatomical model simulates the soft tissues and a plastic resin structure represents the cervical spine bone. An optical sensor was used to measure the displacements performed on simulated skin versus time. The Likert scale was used for assessing the similarity of the anatomical model relative to the size, shape, texture, elasticity and displacement of the skin as well as the curvature of the cervical spine. Five experienced professionals (GP) in the technical performed five series of Pompage technique. With the mean of data collected were determined benchmarks for technical and implemented in a standard guide to train the volunteers. Twenty-six volunteers (GE) with no experience performed the Pompage technique, with the anatomical model following the standard guide. A physical therapist (VE) was selected to evaluate the volunteers (GE) before and after training in the simulator.

ELIGIBILITY:
Inclusion Criteria:

* no history of cervical trauma (GT and VF)
* Do not have dermatitis in the cervical region (GT and VF)
* recurrent migraines (GT and VF)
* no prior knowledge of Pompage technique (GE).
* minimum 5 years experience of applying the Pompage technique (GP and VE).

Exclusion Criteria:

* report pain in the cervical region (GT and VF)
* irritations in the cervical region (GT and VF)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Displacement of the skin | 5 days
  The displacement of the skin (mm) of the volunteers VF and GT was measured to validated the simulator. The volunteers GE used the simulator and the displacement of the skin of simulator was measured during the Pompage technique.
Pressure | 5 days
  The volunteers GE used the simulator and the pressure (mm/Hg ) on the simulator was measured during the Pompage technique.

SECONDARY OUTCOMES:
Cytometry neck | 1 minute
  The cytometry neck (cm) of the volunteers VF and GT was measure to validated the simulator.

CONTACTS AND LOCATIONS:
Overall Officials: Annie F. Frère, PhD, Principal Investigator — University of Mogi das Cruzes

IPD SHARING:
Plan to Share IPD: Yes